CLINICAL TRIAL: NCT05957380
Title: A Multicenter, Double-blind, Active-controlled, Randomized, Parallel Clinical Study to Evaluate the Efficacy and Safety of DA-2803 in Chronic Hepatitis B Patients
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of DA-2803 in Chronic Hepatitis B Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DA2803_HB_IV
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental)
  Interventions: Drug: DA-2803; Drug: Placebo of DA-2803-R
- Reference group (Experimental)
  Interventions: Drug: DA-2803-R; Drug: Placebo of DA-2803

INTERVENTIONS:
Drug: DA-2803 — All participants are administered one tablet per day for 48 weeks
  Arms: Treatment group
Drug: DA-2803-R — All participants are administered one tablet per day for 48 weeks
  Arms: Reference group
Drug: Placebo of DA-2803 — All participants are administered one tablet per day for 48 weeks
  Arms: Reference group
Drug: Placebo of DA-2803-R — All participants are administered one tablet per day for 48 weeks
  Arms: Treatment group

SUMMARY:
This study is a multi-center, double-blind, active-controlled, randomized, parallel clinical study to evaluate the efficacy and safety of DA-2803 in chronic hepatitis B subjects

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects of ages in the range over 19
* The subjects HBsAg positive for at least 6 months or has history of Chronic Hepatitis B
* The subjects whose HBV DNA above 20,000 IU/mL when HBeAg positive or above 2,000 IU/mL when HBeAg negative or positive when has history of Chronic Hepatitis B
* The subjects completely understood the clinical trial through detailed explanation presented, determined to participate in the clinical trial spontaneously, and agreed to observe precautions suggested thereby through written consent

Exclusion Criteria:

* The subjects who have been infected with HCV, HDV, HIV
* The subjects who have Hemochromatosis, Wilson's disease, autoimmune liver disease, and α-1 antitrypsin deficiency
* The subjects whose α-fetoprotein over 50 ng/mL and who are persumed to be Hepatocelluar carcinoma

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
HBV DNA(log10 IU/mL) change | 48 weeks
  HBV DNA(log10 IU/mL) change compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No